CLINICAL TRIAL: NCT05432934
Title: Transversus Abdominis Plane Blocks With and Without Dexamethasone: A Randomized Clinical Trial in Minimally Invasive Colorectal Surgery
Brief Title: Transversus Abdominis Plane Blocks With and Without Dexamethasone
Acronym: TAP-DEX
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Nathan Ginther, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2549
Record Dates: First submitted 2021-09-28; First posted 2022-06-27 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Disorders; Regional Anesthesia Morbidity; Analgesia; Local Anesthetic Complication; Pain, Postoperative; Colorectal Cancer; Crohn Disease; Diverticular Diseases
Keywords: perioperative analgesia; TAP block; laparoscopic surgery; regional anesthesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Colorectal Neoplasms; Crohn Disease; Diverticular Diseases | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 16mg will be added to local anesthetic solution for TAP blocks. 4mg will be injected at 4 anterior abdominal wall sites in a laparoscopically-administered TAP block. This is a single intraoperative dose.
  Interventions: Drug: Dexamethasone
- Local anesthetic only (No Intervention): Local anesthetic (bupivacaine 0.25) 1mL/kg will be used for TAP blocks.

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be added to local anesthetic solution and injected at 4 site for for laparoscopically placed TAP blocks.
  Arms: Dexamethasone

SUMMARY:
Dexamethasone will be used as an adjunct to local anesthetics (bupivacaine) to prolong the duration of laparoscopically-placed transversus-abdominis plane blocks in elective colorectal resection.

DETAILED DESCRIPTION:
Advances in minimally invasive surgery have reduced postoperative morbidity and enhanced recovery. Despite increased use of minimally invasive techniques, postoperative pain remains a challenging aspect of surgical treatment of colorectal diseases and is typically treated with multimodal analgesia, yet the backbone of analgesia continues to be opioid therapy. As analgesics, opioids are effective but fraught with side effects, including delay in return of bowel function, sedation, and potential for dependency.

Minimally invasive colorectal surgery has dramatically improved postoperative outcomes, resulting in significantly shorter length of stay, pain, and overall cost. Despite the advances in multimodal analgesia and enhanced-recovery pathways, the optimal strategy for perioperative analgesia has not yet been defined, and there may be a role for expanded use of regional anesthesia in minimally invasive surgery.

Regional anesthesia, specifically the transversus abdominis plane block, has been shown to reduce postoperative pain and opioid requirements even in the context of minimally invasive surgery. Surgeon-performed, laparoscopically placed TAP blocks are equivalent, or perhaps superior, to ultrasound-guided TAP blocks . Long-acting local anesthetics, specifically liposomal bupivacaine, have been shown to prolong the effect of TAP blocks over non-liposomal bupivacaine , and has also suggested a reduced length of stay and less overall cost, despite the high cost of the formulation. These findings suggest improved outcomes can be expected if a longer block is achieved.

Liposomal bupivacaine is not available and Canada and is very costly. Regional anesthetic supplemented with dexamethasone, a potent corticosteroid, has shown improved efficacy and prolonged duration of anesthetic in other regional anesthetic techniques. The investigators hypothesize that addition of dexamethasone to bupivacaine can prolong the duration of block to be similar to that achieved with liposomal bupivacaine, but at a much lower cost.

Ample evidence exists validating TAP block as an effective adjunct to minimally invasive surgery. Robust data also support the additional benefit of dexamethasone in regional anesthesia. No studies have been published specifically assessing any benefit of combining dexamethasone with local anesthetic to improve the TAP block, and none can be found registered at clinicaltrials.gov. This will be the first such trial to evaluate a promising technique that could reduce postoperative pain and opioid requirements. If found to be effective, this technique would profoundly impact surgical practice around the world.

The investigators propose a multi-centre randomized, single-blinded, controlled trial, enrolling 60 patients. Royal University Hospital in Saskatoon, Saskatchewan will be the primary site, with potential to include at least one additional site. Planning is currently underway to run a second trial site at St. Paul's Hospital, Vancouver, British Columbia. The study investigators maintain a collaborative research relationship with the Division of Colorectal Surgery at the University of British Columbia, and there is potential to leverage this relationship to increase the power and relevance of the trial.

Patients older than 18 years scheduled to undergo elective or urgent inpatient minimally invasive colorectal resection will be recruited. The type and site of extraction incision will be at the surgeon's preference. Exclusion criteria include conversion to laparotomy, perforated viscus, peritonitis, acute diverticulitis, death within 72 hours, and preoperative opioid use. The primary outcome will be total opioid consumption in the first 48 hours after surgery. Secondary outcomes will be time in the PACU and length of stay in hospital. A computer-generated random number table will be used to randomize patients to receive either conventional TAP (n=30) or TAP-DEX (n=30). Allocation will be performed in a 1:1 ratio. Group allocation will be revealed to the operating surgeon in order to administer the correct solution, but blinded to patient and study investigators, PACU staff, and ward staff.

Trial participants will undergo their planned procedures as clinically indicated. Eligible procedures include laparoscopic low anterior resection, anterior resection, and segmental colectomy.

At completion of the surgery, patients will undergo surgeon-placed laparoscopic TAP blocks using 1mL/kg of 0.25% bupivacaine with epinephrine 1:200,000, placed at two locations per side along the anterior axillary line between the costal margin and the iliac crest. The dexamethasone group will have 16mg dexamethasone added to the solution. Intravenous dexamethasone will not be given for prevention of postoperative nausea and vomiting. General anesthetic technique will be at the preference of the anesthesiologist.

Statistical Analysis

Data collection: A blinded, centralized, third-party research assistant will carry out data collection. Postoperative opioid consumption will be quantified through chart review as well as assessment of PCA usage 48 hours following the operation. Recording the doses of opioids administered in the medication administration record (MAR) is standard practice by PACU nursing staff at the study institution. PCA pumps automatically document cumulative opioids administered and can easily be checked at the bedside. Data will be entered and recorded into an encrypted Microsoft Excel spreadsheet.

The study intends to enroll a sample size of 60 patients, with 30 patients in each group, using a power of 80% and alpha set at 5%, to detect a detect a difference of 25% (delta=-0.25) under a normal distribution. Given that the standard deviation of 1 is 0.341 under a normal distribution, the sample size was calculated using a 'power of two means" test with a commercially available software (STATA ®). This same sample size, and power calculation, has been used in several trials before . There is an anticipated reduction from 32mg hydromorphone equivalents in the TAP group to less than 25mg in the TAP-DEX group. Thus, the investigators are confident that enrolling 60 patients will be sufficient to detect at least a 25% difference.

Primary outcome: The primary outcome will be total opioid use, in morphine equivalents, in the post-anesthetic recovery unit and the first 48 hours after surgery, Opioid equivalents will be calculated using http://opioidcalculator.practicalpainmanagement.com/conversion.php.

Secondary Outcome: Secondary outcomes will include time of stay in the PACU and length of stay in hospital.

An interim analysis will be performed after 50% enrolment for evaluation of superiority of either treatment.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* ASA class I-III
* elective or urgent inpatient laparoscopic/laparoscopic assisted colorectal surgery.

Exclusion Criteria:

* emergency surgery
* open surgery
* contraindications to laparoscopic surgery (ie. adhesions, inability to tolerate pneumoperitoneum)
* ASA class 4
* age < 18
* pregnant or breastfeeding women
* significant cardiorespiratory/hepatic/renal disease
* allergy to any study drugs
* inability to consent
* inability to respond to pain assessments
* inability to use the patient-controlled analgesia device (PCA)
* preoperative chronic opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Total postoperative opioid consumption in the first 48 hours after surgery (hydromorphone equivalents. | 48 hours

SECONDARY OUTCOMES:
Opioid consumption in the post-anesthetic care unit (PACU) | 48 hours
  Total opioid consumption during stay in the PACU, measured in hydromorphone equivalents.
Length of stay in post-anesthetic care unit (minutes). | 60-120 minutes
  Total duration of stay in PACU before transfer to the ward, measured in minutes. We anticipate a range of 60-120 minutes.
Length of stay in hospital (days). | 3-7 days
  Total hospital stay, measured in days. Usual range is 3-7 days.

CONTACTS AND LOCATIONS:
Overall Officials: David N Ginther, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT05432934/Prot_000.pdf